CLINICAL TRIAL: NCT01411761
Title: Phase 4 Study of Saccharomyces Boulardii on Indirect Hyperbilirubinemia
Brief Title: Effect of Saccharomyces Boulardii on Indirect Hyperbilirubinemia and Phototherapy Duration in Very Low Birth Weight Infants
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zekai Tahir Burak Women's Health Research and Education Hospital (Other)
Responsible Party: Zekai Tahir Burak Maternity and Teaching Hospital, Zekai Tahir Burak Maternity and Teaching Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: demirel9800
Record Dates: First submitted 2011-08-05; First posted 2011-08-08 (Estimated); Last update posted 2011-08-08 (Estimated); Status verified 2011-06

CONDITIONS: Indirect Hyperbilirubinemia
Keywords: indirect hyperbilirubinemia; very low birth weight infants

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Saccharomyces boulardii (Experimental): study group
  Interventions: Dietary Supplement: Reflor
- placebo (Placebo Comparator): serum physiologic
  Interventions: Other: serum physiologic

INTERVENTIONS:
Dietary Supplement: Reflor — 5 million unit/day, first 15 day of life
  Arms: Saccharomyces boulardii
Other: serum physiologic — 1 cc added to one feeding in a day
  Arms: placebo

SUMMARY:
Indirect hyperbilirubinemia is frequently observed in premature infants.Probiotics are favorable microorganisms that regulate the flora of the gastrointestinal system. In this study we aimed to compare the effect of S. boulardii on severity of hyperbilirubinemia and duration of phototherapy on very low birth weight infants.

ELIGIBILITY:
Inclusion Criteria:

* very low birth weight infants

Exclusion Criteria:

* chromosomal anomalies

Ages: 1 Day to 15 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2011-05; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Effect of S. boulardii on severity of hyperbilirubinemia and phototherapy duration | 6 months

SECONDARY OUTCOMES:
long term effect of S.boulardii on neurodevelopmental outcome | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Gamze Demirel, MD, Principal Investigator — Zekai Tahir Burak Women's Health Research and Education Hospital; Ugur Dilmen, Prof, Study Director — Zekai Tahir Burak Maternit Teaching Hospital
Locations (1):
- Zekai Tahir Burak Maternity Teaching Hospital, Division of Neonatology, Ankara, Turkey (Türkiye)